CLINICAL TRIAL: NCT05813002
Title: Impact of Order of Movement on Nerve Root Function: A Neurophysiological Study With Implications for Neurodynamic Test Sequencing
Brief Title: Impact of Order of Movement on Nerve Root Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Professor-chair of Physiotherapy Department, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: REC-22-06-04-S
Record Dates: First submitted 2023-04-01; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Physical and Rehabilitation Medicine
Keywords: Randomized controlled trial; Neurodynamics; Evoked potential; Somatosensory

STUDY DESIGN:
Intervention Model Description: A prospective, parallel-group, randomized clinical trial participants will be randomly assigned to one of three different groups. One group will receive the standard neural mobilization, the second group will receive Distal-Proximal neural mobilization, and the third group will receive Proximal-Distal neural mobilization, all targeting the median nerve.
Who Masked: Outcomes Assessor
Masking Description: The assessor, who took the measurements for all groups will be blinded to the subject's group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard neurodynamic sequence (Active Comparator): Participants in the first group will receive the standard neurodynamic sequence. The starting position for this sequence will be shoulder in extension with lateral rotation, elbow in full flexion and wrist in neutral position. Passively the shoulder is abducted till 90 degrees followed by wrist extension then ended by elbow extension. Ipsilateral movement of the head bending till 45 degrees with movement of the wrist towards the body for 10 repetitions
  Interventions: Other: standard neural mobilization
- Distal to proximal neurodynamic sequence (Active Comparator): The second group participants will receive the distal to proximal neurodynamic sequence. For this sequence the starting position will be shoulder in full extension with lateral rotation, elbow fully extended and wrist in neutral position. the sequence will start with wrist extension, going to elbow extension, and ending with shoulder abduction. Ipsilateral movement of the head bending till 45 degrees with movement of the wrist towards the body for 10 repetitions
  Interventions: Other: Distal to proximal neural mobilization
- proximal to distal neurodynamic sequence (Active Comparator): The participants in the third experimental group will receive the proximal to distal sequence which will start with shoulder abduction, elbow extension and then wrist extension. The starting position is shoulder in extension and laterally rotated, elbow in full flexion, and wrist in neutral position. The shoulder will be passively mobilized to 90 degrees of abduction, elbow into full extension and wrist in full extension. Ipsilateral movement of the head bending till 45 degrees with movement of the wrist towards the body for 10 repetitions
  Interventions: Other: proximal to distal neural mobilization

INTERVENTIONS:
Other: standard neural mobilization — is a movement-based intervention aimed at restoring the homeostasis in and around the nervous system.
  Arms: standard neurodynamic sequence
Other: Distal to proximal neural mobilization — is a distal to proximal movement-based intervention aimed at restoring the homeostasis in and around the nervous system.
  Arms: Distal to proximal neurodynamic sequence
Other: proximal to distal neural mobilization — is a proximal to distal movement-based intervention aimed at restoring the homeostasis in and around the nervous system.
  Arms: proximal to distal neurodynamic sequence

SUMMARY:
the main objective of this study is to investigate if different neurodynamic test sequencing of the median nerve has a different impact on median nerve root function. We hypothesized that the order of median nerve neurodynamic movements would influence peak-to-peak amplitude and latency.

DETAILED DESCRIPTION:
Neurodynamic concept is used clinically to normalize nerve mobility. It has been manifested in previous studies that neurodynamics have increased mobility by floss like movement of the nerve. Whereas in other studies it has been concluded that neurodynamic techniques has an effect in decreasing fibrous and adhesions between neural tissues and the surrounding tissues therefore giving an outcome of improved infrafasicular gliding.

The upper limb neurodynamic test has an effect to alter the mechanical loads on the nerve by changing its dimensions. For neurodynamic to be more effective, it requires a certain sequence.

The different order of movements will induce different duration of tension in which it will influence the nerve root function, which is needed to be investigated to check for the effectiveness. A previous study has found that the difference of sequence on median nerve, had caused a change on the distribution of the sensory response on the asymptomatic participants. The sensory responses were more prevalent during the neurodynamic of the median nerve when it was applied from a distal to proximal sequence . One of the main purposes of the order of sequences is to add more strain to the nerve segment to increase the sensitivity of the test.

Clinically it has been assumed that the different order of movements could possibly influence the level of strain on a certain nerve segment. When the standard sequence was compared with the distal-to-proximal sequence for the median nerve, there was no physiological difference obtained at the end of the test. In comparison, there was a larger strain in the distal-to-proximal sequence in comparison to the proximal-to-distal sequence observed. However, the longitudinal excursion collected data indicated that the start and end positions for all the three sequences were alike.

In terms of neurophysiological outcomes, in this study we will use the dermatomal somatosensory evoked potential as a primary outcome due to its reliability in comparison with other physiological outcomes. There is a literature gap in regard to the effect of the order of sequence on the median nerve on the nerve root function and this is what the study will focus on. We hypothesized that the order of movements of the median nerve neurodynamic will influence the peak-to-peak amplitude and the latency.

ELIGIBILITY:
Inclusion Criteria:

* not currently experiencing any neck or dominant upper extremity symptoms.
* do not have a history significant for a chronic painful condition.
* do not using pain relievers.

Exclusion Criteria:

* inflammatory joint disease or other systemic pathologies.
* prior history of overt injury and surgery relating to the musculoskeletal system.
* disorder related to the spine and extremities.
* musculoskeletal pain in the last three months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in dermatomal somatosensory evoked potentials. | baseline (pre-treatment) and immediately after the treatment
  In all dermatomes, 2 complete recording runs will be undertaken during each session with averages of 250 to 1200 cortical responses from scalp surface recording electrodes (C3'-C4' in a 10-20 electrode configuration) of the contralateral scalp to the stimulated dermatomes being stimulated. The impedance of ground and scalp electrodes will be maintained at < 5 k Cutaneous areas of C5,C6,C7 sensory roots will be stimulated in lower limb with the electrical impulses of 0.2 ms duration, frequency of 3.3 Hz and intensity 3 times higher than the sensory threshold will be determined individually for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim M moustafa, Professor, Principal Investigator — University of Sharjah

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available to other researchers.